CLINICAL TRIAL: NCT04481074
Title: Effects of Inspiratory Muscle Training in Inspiratory Muscle Endurance, Breathlessness, Inspiratory Muscle Strength, Functional Capacity and Quality of Life in Patients With Interstitial Lung Disease
Brief Title: Inspiratory Muscle Training in Patients With Interstitial Lung Disease
Acronym: IMT-ILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Veronica Franco Parreira, Full Professor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UFMG_IMT-ILD
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Interstitial Fibrosis; Pulmonary Disease; Interstitial Lung Disease; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Pneumonia, Interstitial
Keywords: Inspiratory muscle training; Interstitial lung disease; Inspiratory muscle endurance; Breathless
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases; Lung Diseases, Interstitial; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Dyspnea

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory muscle training group (Experimental): Group intervention: home-based interval inspiratory muscle training during 8 weeks, two sessions with two sets of 30 breaths with one minute rest between them. Load set is determinated weekly, aiming 50% of actual PImax and according to Borg Score.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training will be performed using the tapered flow-resistive loading trainer (POWERbreathe®).

SUMMARY:
The aim of this study is to evaluate the effects of inspiratory muscle training program in inspiratory muscle endurance, breathlessness, inspiratory muscle strength, functional capacity and quality of life in patients with interstitial lung disease. Patients are evaluated before the inspiratory muscle training and after 8 weeks of training.

DETAILED DESCRIPTION:
Inspiratory Muscle Training has been described as an effective intervention and contribute to the improvement of inspiratory muscle function and breathlessness in patients with chronic lung disease. The aim of this study is to evaluate, the effects of inspiratory muscle endurance, breathlessness, inspiratory muscle strength, functional capacity and quality of life in patients with interstitial lung disease. It is a quasi-experimental study. Patients with interstitial lung disease are recruited from interstitial disease ambulatory. In each session patients performs two times 30 breaths with a minute rest between them. The load is set according with 50% of actual PImax, the Borg score should be between 4 and 6, otherwise the load will decrease (if Borg more than 6) or increase (if Borg less than 4). New PImax is measured weekly and the new load is defined following the same protocol for 8 weeks. Patients are evaluated before the inspiratory muscle training and after 8 weeks of training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of interstitial lung disease established by a pulmonologist;
* Absence of clinical exacerbations of the disease in the four weeks prior to the initial data collection;
* Present medical research council scale more than 2;
* Absence of a associated or self reported cardiac, orthopedic and psychiatric diseases,
* Not participating in pulmonary rehabilitation programs;
* Do not use supplemental oxygen therapy while resting.

Exclusion Criteria:

- Inability of the participant to understand or perform the procedures proposed during the evaluations and training program.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Inspiratory muscle endurance | At baseline and after 8 weeks of training
  Endurance time in seconds
Change in Breathlessness | At baseline and after 8 weeks of training
  Medical Research Council (1-5)

SECONDARY OUTCOMES:
Change in Inspiratory muscle strength | At baseline and after 8 weeks of training
  Maximal inspiratory pressure in cmH20
Change in Functional capacity | At baseline and after 8 weeks of training
  Maximal distance in 6 minute walk test
Change in Quality of life | At baseline and after 8 weeks of training
  King's Brief Interstitial Lung Disease Questionnaire. It is a 15 questions questionnaire. Total score can go from 0 - 100, 100 is the better quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Ambulatório Bias Fortes - Ambulatório de Doenças Intersticiais do Hospital das Clínicas da Universidade Federal de Minas Gerais., Belo Horizonte, Minas Gerais
  - Laboratório de Avaliação e Pesquisa em Desempenho Cardiorrespiratório da UFMG, Belo Horizonte, Minas Gerais